CLINICAL TRIAL: NCT00813345
Title: A Role for Light Therapy at Immediate Recovery From Short Duration Ambulatory Anesthesia to Prevent Dysregulation of Circadian Rest-Activity Rhythm in Patients Submitted to Colonoscopy.
Brief Title: Ambulatory Anesthesia and Light Therapy
Acronym: LI-AMB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Direction de la Recherche Clinique et de l'Innovation - Hôpitaux Universitaires de Strasbourg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4057; 2007-A00867-46
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Anesthesia; Colonoscopy
Keywords: anesthesia propofol ambulatory rhythm
MeSH Terms: interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - Light therapy (Experimental): Light therapy (1500 lux)
  Interventions: Other: light therapy (1500 lux)
- B - identical control lamp (Placebo Comparator): identical control lamp
  Interventions: Other: standard light (100 LUX)

INTERVENTIONS:
Other: light therapy (1500 lux) — light therapy (1500 lux) for 90 minutes
  Arms: A - Light therapy
Other: standard light (100 LUX) — standard light (100 LUX) for 90 minutes
  Arms: B - identical control lamp

SUMMARY:
We previously evidenced in both animal models and patients that a short duration ambulatory anesthesia impacts the circadian rest-activity biological rhythm, at least during the first 3 days. The light is the main, natural synchronisateur, of the biological cerebral clock, and is used as therapeutics in chronic disturbances of the circadian rest activity rhythm and of the sleep (Alzheimer disease for example). We would like to test for a simple and safe strategy to prevent such a long-lasting effect of anesthesia on biological clock:the increase of the light intensity at a still physiological level during the initial phase of recovery from anesthesia by using a particular artificial light of color spectrum similar to natural sun daylight.

ELIGIBILITY:
Inclusion Criteria:

* ASA I & II
* ambulatory anesthesia for colonoscopy on Monday or Tuesday
* social security

Exclusion Criteria:

* treatment for cancer
* hypnotics, beta-bloquers
* pregnancy
* legal supervision
* trans 5 meridian travel in the last two months

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Modification of on parametric analysis of circadian rhythm of rest-activity post anesthesia as compared to reference period (within factor) ; between factor : light intensity group | Within the first 5 days after anesthesia

SECONDARY OUTCOMES:
Influence of gene period 3 phenotype on the effect of anesthesia | Blood sample taken the day of the anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Laure PAIN, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (6):
- France (6):
  - Service d'Anestésie et Réanimation - Hôpital Beaujon, Clichy
  - Service d'Anesthésie et Réanimation - Hôpital Pasteur, Colmar
  - Service d'Anesthésie et Réanimation, Hôpital d'Instruction des Armées Legouest, Metz
  - Centre Ambulatoire des Diaconesses, Strasbourg
  - Centre Ambulatoire-Clinique Saint-Odile, Strasbourg
  - Service d'Anesthésie et Réanimation - Hôpital de Hautepierre, Strasbourg